CLINICAL TRIAL: NCT04011579
Title: Multiple Sclerosis Fitness Intervention Training With Pilates Exercises
Brief Title: Pilates Training in Multiple Sclerosis
Acronym: MS-FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Italiana Sclerosi Multipla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FISM 2019MSFIT
Record Dates: First submitted 2019-06-11; First posted 2019-07-08 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis; Physical Activity
Keywords: Physical activity; Pilates; Fitness
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSFIT (Experimental): The MSFIT group will self-manage Pilates exercises at-home through a tool based on XBox Kinect for 12 weeks, performing at least 3 sessions/week for a total of 30 minutes of exercises for each session(also distributed during the day with a minimum slot of 10 minutes). No rehabilitative interventions except sphincter and speech rehabilitation and psychological support, are admitted for the 12 weeks of participation to the project and the following 6 weeks before Follow-up evaluations (a total of 18 weeks). The execution of unspecific physical activities, if not already practiced, will be suggested to the participants.
  Interventions: Other: MSFIT
- CTRL (No Intervention): No rehabilitative interventions except sphincter and speech rehabilitation and psychological support, are admitted for the 12 weeks of participation to the project and the following 6 weeks before Follow-up evaluations (a total of 18 weeks). The execution of unspecific physical activities, if not already practiced, will be suggested to the participants.

INTERVENTIONS:
Other: MSFIT — MSFIT, by using the Microsoft Kinect Motion Controller Xbox to deliver adapted physical activity, offers the possibility to transform the Pilates exercises into a virtual reality game. Each exercise is implemented with different levels of difficulty in order to allow the adaptation to the capacities of the user.
  Arms: MSFIT

SUMMARY:
To date, despite recent advances in MS care including rehabilitation interventions, many PwMS are unable to access these developments due to limited mobility, fatigue and related issues, and costs associated with travel.

Thus, physical activity at home could be a new way to deliver exercises to the patients. Although Pilates did not show any significant advantage over standardized physical therapy in the current literature, it is a good method to promote physical activity, sensorimotor integration and cognitive stimulation. Thus, it could be a treatment option to improve fatigue, balance and walking abilities in PwMS; consequently, Pilates could be suggested by the clinician as a physical activity to be integrated in the daily life.

This possibility could be made more feasible using new tools such as those offered by low cost devices.

The main MS-FIT project purposes are to provide and to test a tool based on serious game concept of Pilates-inspired exercises for daily use at home, by mixing the entertainment aspects typical of the videogames and the possibility to perform physical activity.

The MS-FIT tool does not pursue therapeutic aims as rehabilitation does, but it could have a positive impact on prevention and health in MS.

MS-FIT, by using the Microsoft Kinect Motion Controller Xbox or similar to deliver adapted physical activity, offers the possibility to transform the Pilates exercises into a virtual reality game.

MS-FIT, through a multicentre approach, would provide:

* a feasibility study in order to:

  * refine the tool for the final customized version to be used in a RCT MS study
  * assess the tool for PwMS in terms of technology acceptability and satisfaction-to-use
  * assess the process of recruitment, the adherence to the intervention, the dropout rate and identify potential issues
  * assess human resources necessary for the RCT
  * estimate the effect of the intervention and its variance necessary to calculate the appropriate sample size for the RCT
* a RCT study in order to evaluate the effect of a physical activity intervention of exercises inspired to Pilates self-managed at home in terms on PwMS

DETAILED DESCRIPTION:
Devices and technologies for at-home interventions could provide to PwMS with mild disability useful tools to successfully maintain own physical, cognitive and emotional status by performing at-home physical activity/exercises and avoiding outpatient interventions. Together, new devices and technologies could help in overcoming all barriers (i.e. transportations, working time, etc.) hindering the adherence to and, consequently, efficacy of the outpatient treatments.

Although Pilates did not show any significant advantage over standardized physical therapy in the current literature, it is a good method to promote physical activity, sensorimotor integration and cognitive stimulation. Thus, it could be a treatment option to improve fatigue, balance and walking abilities in PwMS; consequently, Pilates could be suggested by the clinician as a physical activity to be integrated in the daily life.

This possibility could be made more feasible using new tools such as those offered by low cost devices.

The main MS-FIT project purposes are to provide and to test a tool based on serious game concept of Pilates-inspired exercises for daily use at home, by mixing the entertainment aspects typical of the videogames and the possibility to perform physical activity.

The MS-FIT tool does not pursue therapeutic aims as rehabilitation does, but it could have a positive impact on prevention and health in MS.

MS-FIT, by using the Microsoft Kinect Motion Controller Xbox or similar to deliver adapted physical activity, offers the possibility to transform the Pilates exercises into a virtual reality game.

MS-FIT, through a multicentre approach, would provide:

* Feasibility study
* RCT study

All the 14 participating centres will select a dedicated therapist who will be responsible for patient training in using the MS-FIT tool.

All the subjects recruited following the inclusion/exclusion criteria will sign an informed consent and all the procedures (feasibility and RCT) will be in agreement with the Declaration of Helsinki (1964) and approved by Local Ethical Committee.

No trial-specific procedures will be conducted before informed consent has been obtained, and participants will be reminded that they may withdraw from the trial at any time without it affecting the quality of their care in the future.

Participants with relapses during the period of their involvement in the project will be considered as drop out and will be considered in the analysis for the entire period of study participation.

Feasibility study

Primary objective:

• the refinement of the tool for the final customized version to be used in a RCT MS study. The primary objective will be reached by fixing eventual bugs relieved during the feasibility study and taking into account results from the assessment in terms of technology acceptability and satisfaction-to-use, adherence to the intervention, intervention safety and the physical effects of the intervention.

Secondary Objectives:

* the estimation of human resources necessary for the RCT.
* the estimation of the effect of the intervention and its variance necessary to calculate the appropriate sample size for the RCT.

Due to the nature of the feasibility study and based on previous literature showing that a sample size of 25-40 subjects per arm is adequate for a feasibility trial, the investigators will recruit 28 PwMS per arm. All the 14 participating centres will recruit a total of 56 recruited patients following the inclusion and exclusion criteria. In the range of EDSS inclusion criteria 28 subjects will be recruited with lower disability (EDSS 2-3) and 28 with higher disability (EDSS of 3.5 or 4). For both levels the subjects will be randomized into two groups: MSFITFeas (MS-FIT at-home + "unspecific physical activities") and CTRLFeas ("unspecific physical activities"). Randomization will be provided by an independent randomization service at FISM accessed via a web-based system, using computer-based block randomization (1 factor: EDSS score 2-3 and 3.5-4). Patient will be allocated to MSFITFeas and CTRLFeas in a 1:1 ratio. Confirmation emails will be sent to Centres PI.

The MSFITFeas group will self-manage MS-FIT at-home for 6 weeks, performing at least 3 sessions/week for a total of 30 minutes of exercises (also distributed during the day with a minimum slot of 10 minutes) for each session. During this period Xbox One and Microsoft Kinect 2.0 will be delivered to the participants for the aims of the study. Before starting the at-home intervention each subject will be trained to the use of the platform by a therapist. No rehabilitative interventions except sphincter and speech rehabilitation and psychological support, are admitted for the 6 weeks of participation to the project. The execution of unspecific physical activities, if not already practiced, will be suggested to the participants. For the 6 weeks of participation to the project CTRLFeas will be similar to MSFITFeas group except for the execution of MS-FIT at-home.

The protocol for the Feasibility study will consist on (Figure 2):

* T0 evaluation (PRE)
* 6 weeks of intervention

  * MSFITFeas: unspecific physical activities + MS-FIT at-home
  * CTRLFeas: unspecific physical activities
* T1 evaluation (POST)

The evaluation for the Feasibility study are described in the section Outcome Measures.

Deliverables Deliverables of the Feasibility study will be the final customized tool, a set of indications for the management of the RCT, the sample size estimation for the RCT.

Focus group A nested qualitative study on 14 participants will explore patients' experiences of MS-FIT via Focus Group Meeting (FGM). The objectives are to provide insight into the quantitative results, explore strengths and limitations of the intervention with MS-FIT, so as to guide the RCT.

The report of each FGM analysis will be submitted to FGM participants for review (respondent validation).

Deliverables Deliverables of the nested qualitative study will be the delivery of the report of the FGM analysis.

RCT study

Primary Objective:

• evaluation of the change in TUG.

Secondary Objectives:

* evaluation of the physical effects also in terms of self-reported outcome, upper limb performances, resistance in walking and physical activity, cognitive and psychosocial effects, quality of life and wellbeing. Differences in physical and cognitive performances due to the genetic features will be evaluated also considering subgroups identified through the polymorphism analysis.
* evaluation of the acceptability and satisfaction-to-use, adherence to the intervention, intervention safety through the measurements of endpoint already listed for the Feasibility study.

The RCT sample size will be definitively calculated based on the results from the feasibility study. However, by considering the literature about Pilates in MS, the investigators can preliminary estimate the needed sample size. In particular, the investigators refer to the TUG post-intervention improvement found by Karlon et al. in a group of PwMS performing Pilates. For our aim, the investigators can consider this result even if no differences between Pilates group and control group (Physiotherapy) were found. Pilates group improved the performance in TUG of about 1.8s, that could be considered as clinically relevant for PwMS. By considering a variability of about 3.4s, a power of 80%, a level of significance (two sided) of 5% and a potential loss of 15% of patients at follow-up, the estimation of the necessary sample size consists of approximately 63 subjects for the experimental group (a total of 126).

All the 14 participating centres will be involved in the patients' enrolment. The subjects will be randomized into two groups: MSFITRCT (MS-FIT at-home + "unspecific physical activities") and CTRLRCT ("unspecific physical activities"). The randomization will be carried out using a web based procedure and will be centrally managed. A stratified minimization/adaptive algorithm will be used in order to balance the baseline EDSS (2-3 vs 3.5-4) factors across the two groups.

The MSFITRCT group will self-manage MS-FIT at-home for 12 weeks, performing at least 3 sessions/week for a total of 30 minutes of exercises (also distributed during the day with a minimum slot of 10 minutes) for each session. During this period Xbox One and Microsoft Kinect 2.0 will be delivered to the participants for the aims of the study. Before starting the at-home intervention each subject will be trained to the use of the platform by a therapist. The follow-up (FU) evaluation will be after 6 weeks since the end of the intervention. No rehabilitative interventions except sphincter and speech rehabilitation and psychological support, are admitted for the 18 (12 + 6) weeks of participation to the project. The execution of unspecific physical activities, if not already practiced, will be suggested to the participants. For the 18 (12 + 6) weeks of participation to the project CTRLFeas will be similar to MSFITFeas group except for the execution of MS-FIT at-home.

At the end of the 18 weeks, the participants of the CTRLRCT group will be offered the MS-FIT intervention.

The requirement that the enrolled patients will have not to perform any supervised physical activity or rehabilitative intervention is in line with recent studies showing that most of PwMS with mild disability (78.34% EDSS <4) were not treated with rehabilitation.

The subjects involved in the feasibility study will be excluded from the RCT study in order to avoid bias effects.

The protocol design for the RCT study will consist on (Figure 3):

* T0 evaluation (PRE)
* 12 weeks of intervention

  * MSFITRCT: unspecific physical activities + MS-FIT at-home
  * CTRLRCT: unspecific physical activities
* T1 evaluation (POST)
* T2 evaluation (FU) - after 6 weeks from T1

The evaluation for the RCT study are described in the section Outcome Measures. Moreover, blood samples will be collected at T0 to investigate if genetic polymorphisms of candidate regulators of neuronal plasticity could be correlated to the response to the proposed protocol. According to previous report MS subjects of the two RCT groups could be subdivided in subgroups with respect to the polymorphism features. For example, for the CNR1 gene the subdivision could be based on the number of AAT repetitions (short AAT: homozygous or heterozygous for allele with ≤11 repeats of AAT triplets; long AAT: homozygous for allele with ≥12 repeats of AAT triplets).

Differences among subgroups in terms of physical and cognitive performances will be evaluated.

In particular, all patients will be genotyped for a total of 55 genetic polymorphisms of 23 potential regulators, like: Homer1; AKT1; RAPTOR; D2R; GAPD; CHAT; p53; BRCA2; LIG4; XRCC5; CYP3A4; NBS1; MDM2; CNR1, ATTn; CNR2; GRIN1; GRIN2B; TRPV1; FAAH, COMPT; (Brain-derived neurotrophic factor) BDNF.

Blood sample will be assessed from participants early in the morning after awakening (8h). To synchronize the sample for lifestyle variables, subjects were requested to avoid excessive physical activity the last three days before the blood sampling, sleep for 7-8h the night before study, avoid starving, and eat a usual breakfast in the morning (approximately 1h before the time of the breakfast).

The samples will be collected by each participant centre and shipped to the IRCCS Neuromed, Pozzilli, Isernia (Prof. Diego Centonze) for the analyses.

Deliverables Deliverables will be the report of the results of the trial and the final guidelines to make available and easy-to-use the MS-FIT tool

Criteria for Premature Withdrawal

Criteria for the premature withdrawal are:

1. Patients withdrawal of the consent anytime;
2. Any medical conditions that the investigator determines jeopardize the patient's safety if she/he continues the study and/or study results;
3. Patient's no-compliance to complete the study procedures
4. MS Treatment changes during the study

ELIGIBILITY:
Inclusion Criteria:

* All disease courses of MS
* Expanded Disability Status Scale (EDSS) 2-4
* Hospital Anxiety and Depression Scale (HADS) < 10 in the two subset of anxiety and depression
* Berg Balance Scale (BBS) > 46
* Mini-Mental State Examination (MMSE) > 24
* At least 1 month without having been treated with rehabilitation
* Willingness to sign informed consent

Exclusion Criteria:

* Visual deficits that could compromise the use of MS-FIT
* Relapses in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Change in Timed Up & Go (TUG) | T0: before intervention; T1: after 12 weeks of intervention; T2: 6 weeks after T1
  The Timed "Up and Go" Test measures, in seconds, the time taken by an individual to stand up from a standard arm chair (approximate seat height of 46 cm, arm height 65 cm), walk a distance of 3 meters (approximately 10 feet), turn, walk back to the chair, and sit down.

SECONDARY OUTCOMES:
Change in Timed 25-Foot Walk (T25FW) | T0: before intervention; T1: after 12 weeks of intervention; T2: 6 weeks after T1
  The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk.The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk.
Change in Ambulation Index (AI) | T0: before intervention; T1: after 12 weeks of intervention; T2: 6 weeks after T1
  The AI is a rating scale developed by Hauser et al (1983) to assess mobility by evaluating the time and degree of assistance required to walk 25 feet. Scores range from 0 (asymptomatic and fully active) to 10 (bedridden). The patient is asked to walk a marked 25-foot course as quickly and safely as possible. The examiner records the time and type of assistance (e.g., cane, walker, crutches) needed.
Change in 2-Minutes Walking Test (2WT) | T0: before intervention; T1: after 12 weeks of intervention; T2: 6 weeks after T1
  The 2-minute walk test (2WT) is an easy to perform and practical test that has been used in the assessment of patients with a variety of diseases. It simply measures the distance that a patient can walk on a flat, hard surface in a period of 2 minutes.
Change in Technology Acceptance Model (TAM) | T0: before intervention; T1: after 12 weeks of intervention; T2: 6 weeks after T1
  The technology acceptance model (TAM) is an information systems theory that models how users come to accept and use a technology. The model suggests that when users are presented with a new technology, a number of factors influence their decision about how and when they will use it, notably: the Perceived usefulness and the Perceived ease-of-use.
Change in Client Satisfaction Questionnaire-8 (CSQ-8) | T0: before intervention; T1: after 12 weeks of intervention; T2: 6 weeks after T1
  The CSQ-8 is the most used self-report questionnaires constructed to measure satisfaction with services received by individuals and families. The item score ranges from 1 to 4 and the maximum total score is 32. Higher values mean met needs.
Change in Telehealth Satisfaction Scale (TeSS) | T0: before intervention; T1: after 12 weeks of intervention; T2: 6 weeks after T1
  Evaluation of the level of satisfaction with telehealth from the perspective of clinic patients.The item score ranges from 1 to 4 and the maximum total score is 40. Higher values mean excellent satisfaction.
Adherence to the intervention based on sessions | T1: after 12 weeks of intervention
  Number of sessions actually performed
Adherence to the intervention based on drop-out | T1: after 12 weeks of intervention
  Number of dropout
Change in Twelve Item MS Walking Scale (MSWS-12) | T0: before intervention; T1: after 12 weeks of intervention; T2: 6 weeks after T1
  The 12-item Multiple Sclerosis Walking Scale (MSWS-12) is a self-report measure of the impact of MS on the individual's walking ability. The item score ranges from 1 to 5 and the maximum total score is 60. Lower values mean lower disease impact on walking.
Change in Visual Analogue Scale (VAS) (0-10) for balance performance | T0: before intervention; T1: after 12 weeks of intervention; T2: 6 weeks after T1
  Balance performance subjective evaluation on a scale of 10 points. Subjects have to indicate the self-perceived balance performance in a line ranging from 0 to 10.
Change in Nine-Hole Peg Test (9HPT) | T0: before intervention; T1: after 12 weeks of intervention; T2: 6 weeks after T1
  The Nine-Hole Peg Test (9HPT) is a test used to measure finger dexterity in patients with various neurological diagnoses.
Change in Modified Fatigue Impact Scale (MFIS) | T0: before intervention; T1: after 12 weeks of intervention; T2: 6 weeks after T1
  MFIS is a 21-items questionnaire and provides a subjective assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The item score ranges from 0 to 4 and the maximum total score is 84. Lower values mean lower self-perceived effect of fatigue. Physical subtest range from 0 to 36. Cognitive subtest ranges from 0 to 40. Psychosocial subtest ranges from 0 to 8.
Change in Brief International Cognitive Assessment for MS (BICAMS) | T0: before intervention; T1: after 12 weeks of intervention; T2: 6 weeks after T1
  The Brief International Cognitive Assessment for MS (BICAMS) battery includes Symbol Digit Modality Test (SDMT) for information processing, Californian Verbal Learning Test (CVLT) for verbal memory, Visuospatial Memory Test (BVMT) for spatial memory. In SDMT subjects have to assign as fast and as accurate as possible the numbers 1-9 to predefined symbols in 90s. In VLMT the examiner reads aloud and consecutively the 15 words to the participant who in return has to recall as many words as possible. This procedure is repeated 5 times. The sum score is the number of correctly recalled words. In BVMT subjects have to encode 6 geometrical figures and memorize their precise location during presentation of 10s. Immediately afterwards, subjects have to draw the memorized figures in the right location. The procedure is repeated 3 times. Depending on figure and exact location accuracy, a scoring from 0 to 2 points for each figure is given. The total recall score is the sum of the three trials.
Change in Patient Global Impression of Change (PGIC) with a 7-points scale | T1: after 12 weeks of intervention; T2: 6 weeks after T1
  The self-report measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment. PGIC is a 7 point scale depicting a patient's rating of overall improvement. It has the options "very much improved", "much improved", "minimally improved", "no change", "minimally worsened", "much worsened", and "very much worsened".
Change in Multiple Sclerosis Quality of Life-54 (MSQoL54) | T0: before intervention; T1: after 12 weeks of intervention; T2: 6 weeks after T1
  The MSQOL-54 is a multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument. There is no single overall score for the MSQOL-54. Two summary scores - physical health and mental health - can be derived from a weighted combination of scale scores. In addition, there are 12 subscales: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function. There are also two single-item measures: satisfaction with sexual function and change in health. See the original article describing the development and testing of the MSQOL-54 (Vickrey et al, 1995) for details. Administration forms and scoring instructions can be downloaded.
Change in Psychological Well-Being Scales (PWB) | T0: before intervention; T1: after 12 weeks of intervention; T2: 6 weeks after T1
  PWB measures 6 aspects of wellbeing/happiness that respondents rate statements on a scale of 1 to 6, with 1 indicating strong disagreement and 6 indicating strong agreement.
  Self-acceptance: High scorer: Possesses a positive attitude toward the self; Low scorer: Feels dissatisfied with self.
  Positive relations with others: Higher score: Has warm, satisfying, trusting relationships with others; Lower score: Has few close, trusting relationships with others.
  Autonomy: High scorer: Is self-determining and independent; Low scorer: Is concerned about the expectations and evaluations of others.
  Environmental mastery: High scorer: Has a sense of mastery and competence in managing the environment; Low scorer: Has difficulty managing everyday affairs; Purpose in life: High scorer: Has goals in life and a sense of directedness; Low scorer: Lacks a sense of meaning in life.
  Personal growth: High scorer: Has a continued development feeling; Low scorer: Has a personal stagnation sense.
Change in International Physical Activity Questionnaire (IPAQ) | T0: before intervention; T1: after 12 weeks of intervention; T2: 6 weeks after T1
  IPAQ is a method for physical activity assessment of time spent in several domains. In particular 5 domains are considered: JOB-RELATED; TRANSPORTATION; HOUSEWORK, HOUSE MAINTENANCE, AND CARING FOR FAMILY; RECREATION, SPORT, AND LEISURE-TIME; TIME SPENT SITTING.
  Three levels of physical activity are proposed:
  Low: Those individuals who not meet criteria for categories 2 or 3.
  Moderate:
  * 3 or more days of vigorous activity of at least 20 minutes per day
  * 5 or more days of moderate-intensity activity or walking of at least 30 minutes per day
  * 5 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 600 (metabolic equivalent)MET-min/week.
  High:
  * Vigorous-intensity activity on at least 3 days and accumulating at least 1500 MET-minutes/ week OR
  * 7 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 3000 MET-minutes/week.
Change in Minnesota Leisure-Time Physical Activity Questionnaire | T0: before intervention; T1: after 12 weeks of intervention; T2: 6 weeks after T1
  Assessment of physical activity in terms of total energy expenditure. The results were expressed in a weekly value [kcal/week] after dividing the calcu- lated 6-month energy expenditure by 26 weeks. The following ranges of activity intensity were used: low [< 4 MET], medium [4 - < 6 MET] and high [≥ 6 MET], where 1 MET equals the resting metabolic rate, which is approximately 3.5 ml oxygen kg-1 body weight per min-1.
Correlation between genetic polymorphisms and response to protocol | T0: before intervention
  Blood samples at baseline to genotype the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Giampaolo Brichetto, Principal Investigator — Italian Multiple Sclerosis Foundation
Locations (1):
- Italian Multiple Sclerosis Foundation, Genoa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tacchino A, Ponzio M, Confalonieri P, Leocani L, Inglese M, Centonze D, Cocco E, Gallo P, Paolicelli D, Rovaris M, Sabattini L, Tedeschi G, Prosperini L, Patti F, Sessa E, Pedrazzoli E, Battaglia MA, Brichetto G. Effect of an Internet-Based Pilates Telerehabilitation Intervention in People With Multiple Sclerosis: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Feb 3;14:e58026. doi: 10.2196/58026. PMID 39899835